CLINICAL TRIAL: NCT00166933
Title: Minimal Erythema Dose of UV-B in Normal Population of Taiwan
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700530
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-08

CONDITIONS: Human Volunteers
Keywords: minimal erythema dose; UVB; normal

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
There is no previous study on the minimal erythema dose of UVB irradiation in Chinese people. We will investigate the correlation of skin phototype, constitutive skin color, facultative skin color and minimal erythema dose in Taiwanese.

DETAILED DESCRIPTION:
The skin phototype will be obtained from a structuralized questionaire. The constitutive skin color and facultative skin color will be obtained by chromameter. The minimal erythema dose will be obtained by physician's assessment.

ELIGIBILITY:
Inclusion Criteria:

10-65 years old normal healthy volunteers

Exclusion Criteria:

Age under 10 years old or older than 65 years old People with a past history of photo-sensitivity People who had been treated with phototherapy

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, MD, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- Chia-Yu Chu, Taipei, Taiwan